CLINICAL TRIAL: NCT02482753
Title: A Phase III Trial of Chidamide in Combination With Exemestane in Patients With Hormone Receptor-Positive Advanced Breast Cancer (ACE)
Brief Title: Trial of Chidamide in Combination With Exemestane in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDM301
Record Dates: First submitted 2015-06-17; First posted 2015-06-26 (Estimated); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
Keywords: Chidamide; breast cancer; exemestane; Estrogen Receptor
MeSH Terms: conditions — Breast Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; exemestane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Chidamide + exemestane, open-label (Experimental): Patients receive 30 mg Chidamide per week and 25 mg exemestane QD. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Chidamide; Drug: exemestane
- Chidamide + exemestane, double-blinded (Experimental): Patients receive 30 mg Chidamide twice per week and 25 mg exemestane QD. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Chidamide; Drug: exemestane
- placebo + exemestane, double-blinded (Placebo Comparator): Patients receive placebo twice per week and 25 mg exemestane PO QD. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: exemestane; Drug: placebo

INTERVENTIONS:
Drug: Chidamide — 30 mg, administered orally twice per week (BIW)
  Other Names: CS055
  Arms: Chidamide + exemestane, double-blinded; Chidamide + exemestane, open-label
Drug: exemestane — 25 mg, PO daily
  Other Names: Aromasin
Drug: placebo — Administered orally twice per week (BIW)
  Other Names: Simulation tablet of Chidamide
  Arms: placebo + exemestane, double-blinded

SUMMARY:
This study was to evaluate the efficacy and safety of Chidamide in combination with exemestane in postmenopausal patients with hormone-receptor positive advanced breast cancer.

DETAILED DESCRIPTION:
This study including two parts: (1) Part A, open-label design, 20 patients will be enrolled and receive 30 mg Chidamide BIW and 25 mg exemestane QD. The main object of part A is to evaluate the pharmacokinetic and pharmacodynamic profile of Chidamide when in combination with exemestane. (2) Part B, randomized and double-blinded design, 328 patients will be assigned randomly in a 2:1 ratio to experiment group (30 mg Chidamide BIW + 25 mg exemestane QD) and control group (placebo BIW + 25 mg exemestane QD), to evaluate the efficacy and safety of Chidamide when in combination with exemestane in patients with locally advanced or metastatic estrogen receptor-positive breast cancer progressing on endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ~ 75 years old, postmenopausal women;
2. Histological or cytological confirmation of hormone receptor-positive [estrogen receptor (ER) positive and progesterone receptors (PgR) positive or negative] breast cancer;
3. Disease progression or recurrence after at least one endocrine therapy (either in advanced/metastatic setting or adjuvant setting);
4. ≤4 prior therapies (either in advanced/metastatic setting or adjuvant setting), patients may have received one prior chemotherapy;
5. The disease condition is inoperable, stage III or stage IV, at least one measurable lesion or simple bone metastases with no measurable lesions;
6. Last prior therapy intervals: (a) if the last treatment was endocrine therapy, the interval must ≥ 2 weeks; (b) if the last treatment was chemotherapy therapy, the interval must ≥ 4 weeks;
7. Eastern Cooperative Oncology Group Performance Status: 0~1;
8. Absolute neutrophil count ≥ 1.5×109 / L, platelet count ≥ 100×109 / L, hemoglobin ≥ 90 g/L;
9. Life expectancy ≥ 3 months;
10. Have signed informed consent.

Exclusion Criteria:

1. Patients have known central nervous system (CNS) metastases or a history of CNS metastases , or with leptomeningeal disease;
2. Patients with human epidermal growth factor receptor-2 (Her-2) positive;
3. Patients previously received treatment with exemestane;
4. Patients received radiotherapy ≤ 4 weeks prior to study entry;
5. Patients with no measurable lesion (except simple bone metastasis), such as pleural or pericardial effusion, ascites, et al;
6. Patients have uncontrolled or significant cardiovascular disease, including:

   1. Myocardial infarction (< the last 12 months)
   2. Uncontrolled angina (< the last 6 months)
   3. Congestive heart failure (< the last 6 months), or Left Ventricular Ejection Fraction (LVEF) < 50% prior to study entry
   4. History of any significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or TdP)
   5. History of significant QT interval prolongation, or Corrected QT Interval (QTc) > 450 ms prior to study entry
   6. History of cerebrovascular accident
   7. Symptomatic coronary heart disease requiring treatment with agents
7. The size of fluid area detected by cardiac ultrasonography in cavum pericardium is ≥10mm during diastolic period;
8. History of organ transplantation;
9. Patients have not recovered from all clinically relevant toxicities to grade 1 due to prior therapies;
10. Patients have clinical significant gastrointestinal abnormality, e.g., unable to swallow, chronic diarrhea, ileus, that would interfere the ingestion,transportation or absorption of oral agents;
11. Active infection [Suffered from active infection of bacteria, virus, fungi, mycobacteria, parasites, or other infections (excluding nail bed fungal infections), or require intravenous antibiotic therapy, or antiviral therapy, or hospitalization due to any significant infection events], or persistent fever within 14 days prior to study entry;
12. Patients had organ surgery < 6 weeks prior to study entry;
13. Abnormal liver function [total bilirubin > 1.5×upper limit of normal (> 3×upper limit of normal in case of Gilbert syndrome); Transaminases (ALT, AST) >2.5×upper limit of normal (>5x upper limit of normal patients with liver metastases), abnormal renal function (serum creatinine > 1.5×upper limit of normal);
14. Patients with prior invasive malignancies with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ, unless received curative treatment and with documented evidence of no recurrence in the past five years;
15. Any mental or cognitive disorder, that would interfere the ability to understand the informed consent document or the operation and compliance of study;
16. Patients are currently enrolled in another investigational drug study, or completed within 4 weeks prior to study entry, with the exception of patients only in overall survival follow-up;
17. Any other condition which is inappropriate for the study in the opinion of the investigators.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS), double-blinded period | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  PFS is measured from the date of randomization until progression or death, whichever is first met
pharmacokinetic profiles of Chidamide, open-label period | 0,1,2,4,8,12,24,48,72 hours after the first dose of Chidamide on day 2 at induced stage (4 days in total); 0,1,2,4,8,12,24,48,72 hours post-dose on day 1 of cycle 1 at combination treatment stage
  The pharmacokinetic parameters include Area under the plasma concentration versus time curve (AUC) , Peak Plasma Concentration (Cmax), time to reach Cmax (Tmax), mean concentration at steady state (Css)
pharmacokinetic profiles of exemestane, open-label period | 0,1,2,4,8,12,24 hours after the first dose of exemestane on day 1 at induced stage (4 days in total); 0,1,2,4,8,12,24,48,72 hours post-dose on day 1 of cycle 1 at combination treatment stage
  The pharmacokinetic parameters include Area under the plasma concentration versus time curve (AUC) , Peak Plasma Concentration (Cmax), time to reach Cmax (Tmax), mean concentration at steady state (Css)
acetylation level of histone H3, open-label period | pre-dose of Chidamide on day 2 at induced stage (4 days in total); pre-dose of Chidamide on day 1 of cycle 2 at combination treatment stage
  The acetylation level of histone H3 is assayed by enzyme-linked immuno sorbent assay (ELISA).

SECONDARY OUTCOMES:
overall survival, double-blinded period | Time from randomization to death from any cause, assessed up to 6 years
  OS is measured from the date of randomization until death
duration of response (DOR), double-blinded period | From the first date of response until the date of first documented progression, assessed up to 3years
  DOR is measured from the first date when criteria for response is met until the first date when the criteria for progression is met
objective response rate (ORR), open-label period and double-blinded period | Response is assessed once every 6 weeks, assessed up to 3 years
  ORR is defined as percentage of participants with Complete Response and Partial Response, assessed by the investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST)
clinical benefit rate (CBR), open-label period and double-blinded period | Response is assessed once every 6 weeks, assessed up to 3 years
  ORR is defined as percentage of participants with Complete Response, Partial Response or Stable Disease ≥ 24 weeks, assessed by the investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST)
PFS, open-label period | Time from the start of treatment to the earliest of documented disease progression, or death, assessed up to 3 years
  PFS is measured from the start of treatment until progression or death, whichever is first met

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, Principal Investigator — 307 Hospital of PLA
Locations (22):
- China (22):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The 307th Hospital of Chinese people's Liberation Army, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Tumor Hospital of Hebei Province, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Zhejiang Cancer Hospital, Hangzhou, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University ZhongShan Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang Z, Li W, Hu X, Zhang Q, Sun T, Cui S, Wang S, Ouyang Q, Yin Y, Geng C, Tong Z, Cheng Y, Pan Y, Sun Y, Wang H, Ouyang T, Gu K, Feng J, Wang X, Wang S, Liu T, Gao J, Cristofanilli M, Ning Z, Lu X. Tucidinostat plus exemestane for postmenopausal patients with advanced, hormone receptor-positive breast cancer (ACE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Jun;20(6):806-815. doi: 10.1016/S1470-2045(19)30164-0. Epub 2019 Apr 27. PMID 31036468